# ADAPTATION OF COMMUNITY REINFORCEMENT APPROACH FOR THE TREATMENT OF DRUG ADDICTION



**MUHAMMAD SAGHIR** 

DR. MAZHAR IQBAL BHATTI

74-FSS/PHDPSY/F-18

Associate Professor (supervisor)

**Department of Psychology** 

**Faculty of Social Sciences** 

**International Islamic University Islamabad** 

July 10, 2024

### Statistical Analysis Plan

The collected data for this clinical trial was analyzed using SPSS 25 version. Important statistical analysis includes independent sample t-test, paired sample t-tests and one way ANOVA was used. Following are the defining parameters.

## **Independent sample t-test**

Independent sample t-test was used to understand the efficacy of the treatment program between control and experimental groups.

### Paired sample t-test

Paired sample t-test was used to elaborate the differences between the level of assessment. In order to assess the differences on pre and post assessment of interventions based on SCL-90 (scale of comorbidity).

# One way ANOVA

One way ANOVA was used to understand the differences between pre assessment, post assessment and follow up to draw conclusion about the recovery of the participants which is measured by ARQ (Addiction recovery questionnaire).